CLINICAL TRIAL: NCT01477125
Title: Computerised Working Memory Training in Adults With ADHD: A Randomised Controlled Trial
Brief Title: Working Memory Training in Adults With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Swedish Prison and Probation Services (Unknown); The Söderströmska-Königska Foundation (Unknown)
Responsible Party: Principal Investigator, Ylva Ginsberg, MD, PhD, Senior consultant psychiatrist, clinical postdoc, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X002; DAT-NSP (Other: Karolinska Institutet); DAT-KV (Other: Karolinska Institutet)
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: adhd; adults; working memory; training; RCT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flex working memory training (Experimental): 30-40 minutes of working memory training, 5 days a week for 5 weeks
  Interventions: Behavioral: Flex working memory training
- Control version of Flex (Placebo Comparator): 30-40 minutes of training with a control version of Flex, 5 days a week for 5 weeks.
  Interventions: Behavioral: Flex working memory training

INTERVENTIONS:
Behavioral: Flex working memory training — 30-40 minutes of working memory training, 5 days a week for 5 weeks

SUMMARY:
The purpose of this study is to evaluate whether computerised working memory training improves cognitive performance, ADHD symptoms, psychosocial functioning and quality of life in adults with ADHD, from psychiatric outpatient clinics (N=100) as well as from a high-security prison facility (N=50).

DETAILED DESCRIPTION:
The primary aim is to evaluate whether 5 weeks of computerised working memory training improves working memory capacity. Secondary aims are to explore whether improvements in working memory capacity will be transferred to improvements in learning abilities and fluid intelligence. Also, far transfer effects on executive functioning, ADHD symptoms, psychosocial functioning and quality of life will be explored. Finally, it will also be assessed to what extent improvements gained from 5 weeks of working memory training will be maintained 3 and 6 months post-study, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ADHD according to DSM-IV criteria; ADHD combined type, ADHD inattentive type or ADHD UNS, primarily inattentive type.
* Unmedicated for ADHD during the course of the trial, or being under stable ADHD medication for at least one month at baseline visit and without any planned changes in medication until post-study assessments have taken place.

Exclusion Criteria:

* Previous participation in computerised working memory training (completed training).
* Any psychiatric disorder that in the judgment of the investigator, may interfere with study participation and/or study assessments, also including current substance abuse.
* Participation in psychological treatment addressing ADHD during the course of the 5-week training period (psychoeducation is accepted).
* Initiation of psychological treatment for coexistent disorders during the course of the study (treatment already ongoing at baseline visit is accepted if there are no planned changes during the 5-week training period).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-11; Primary Completion 2017-12-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change in a composite measure of working memory capacity | Baseline and 7 weeks
  The composite measure of working memory capacity comprises the sum score of:
  * Digit Span score (forwards/backwards)
  * Span Board score (forwards/backwards)
  * Arithmetics score
  * Spatial Working Memory score

SECONDARY OUTCOMES:
Change in a composite measure of working memory capacity | Baseline and 31 weeks
  The composite measure of working memory capacity will be assessed in a 6-month follow-up conducted at week 31 post-baseline, equivalent to week 24 post-intervention, to assess retention of any training-related improvements.
Change in Digit Span Forwards/Backwards score | Baseline, 7 and 31 weeks
  Evaluating changes in both Digit Span forwards and backwards scores, as measures of simple verbal working memory capacity.
Change in Span Board Forwards/Backwards score | Baseline, 7 and 31 weeks
  Evaluating changes in both Span Board forwards and backwards scores as measures of simple visuo-spatial working memory capacity.
Change in Arithmetics score | Baseline, 7 and 31 weeks
  Evaluating change in Arithmetics score, as a measure of complex verbal working memory capacity as well as of mathematics ability.
Change in Spatial Working Memory score | Baseline, 7 and 31 weeks
  Evaluating change in Spatial Working Memory score as a measure of complex visuo-spatial working memory capacity.
Change in Qbtest scores | Baseline, 7 and 31 weeks
  Evaluating changes in Qbtest, a computerised CPT that in addition to measuring inattention and impulsivity also captures motor activity by an IR device during performance of the CPT.
Change in Raven´s Standard Progressive Matrices score | Baseline, 7 and 31 weeks
  Evaluating change in score of a short version of Raven´s Standard Progressive Matrices, as a measure of fluid intelligence.
Change in Adult ADHD Self-Report Scale (ASRS-v1.1) Symptom Checklist | Baseline, 7, 19, and 31 weeks
  Evaluating changes in ADHD symptoms by self-reported and informant-reported (significant other) versions of ASRS-v1.1, conducted at baseline, post-intervention, at 3-month and 6-month follow-up.
Change in Sheehan Disability Scale (SDS) | Baseline, 7, 19, and 31 weeks
  Evaluating changes in psychosocial functioning by the self-reported SDS conducted at baseline, post-intervention, at 3-month and 6-month follow-up.
Change in EuroQol- 5 Dimensions (EQ-5D) questionnaire | Baseline, 7, 19, and 31 weeks
  Evaluating change in health-related quality of life by the self-reported generic QoL questionnaire EQ-5D, conducted at baseline, post-intervention, at 3-month and 6-month follow-up.
Change in Adult ADHD Quality of Life Measure (AAQoL) | Baseline, 7, 19, and 31 weeks
  Evaluating change in health-related quality of life by the self-reported ADHD specific QoL measure AAQoL, conducted at baseline, post-intervention, at 3-month and 6-month follow-up.
Montgomery Åsberg Depression Rating Scale-Self report (MADRS-S) | Baseline and 7 weeks
  Evaluating if depressive symptoms during the training period, as measured by the self-reported MADRS-S will influence adherence to and results of the working memory training.
Adverse events | Baseline and 7 weeks
  All adverse events that occurred during the course of the 5-week intervention will be collected as part of the post-intervention assessments at week 7.

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Ginsberg, MD, PhD, Principal Investigator — Karolinska Institutet; Henrik Larsson, PhD, Study Director — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden